CLINICAL TRIAL: NCT04073797
Title: PET Imaging of Inflammation and Lipid Lowering Study
Acronym: PIILL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Wellcome Trust (Other); GE Healthcare (Industry); Lund University (Other)
Responsible Party: Principal Investigator, Jason Tarkin, Wellcome Clinical Research Career Development Fellow & Honorary Consultant Cardiologist, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: A095007 (PIILL)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hypercholesterolemia; Hypercholesterolemia, Familial; Atherosclerosis; Carotid Artery Plaque
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II; Atherosclerosis; Carotid Stenosis | interventions — ALN-PCS; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable CVD - treatment (Experimental): Stable CVD with LDL ≥2.6 despite maximally tolerated statins ± other lipid lowering therapies, randomised to add on therapy with inclisiran + placebo tablet
  Interventions: Drug: Inclisiran; Diagnostic Test: 68Ga-DOTATATE PET-MRI
- Stable CVD - placebo control (Active Comparator): Stable CVD with LDL ≥2.6 despite maximally tolerated statins ± other lipid lowering therapies, randomised to placebo injection + colchicine tablet
  Interventions: Diagnostic Test: 68Ga-DOTATATE PET-MRI; Drug: Colchicine
- HeFH - treatment (Placebo Comparator): Stable CVD with LDL ≥2.6 despite maximally tolerated statins ± other lipid lowering therapies, randomised to placebo injection + placebo tablet
  Interventions: Drug: Inclisiran; Diagnostic Test: 68Ga-DOTATATE PET-MRI

INTERVENTIONS:
Drug: Inclisiran — Inclisiran 284 mg, one injection
  Arms: HeFH - treatment; Stable CVD - treatment
Diagnostic Test: 68Ga-DOTATATE PET-MRI — 68Ga-DOTATATE PET-MRI at baseline and 12 weeks
Drug: Colchicine — Colchicine 500 mcg tablet once daily
  Arms: Stable CVD - placebo control

SUMMARY:
While 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) imaging has been used as an early marker of drug efficacy in numerous clinical cardiovascular drug trials, as a glucose analog, its signal in the vasculature lacks inflammatory cell-specificity. Moreover, high background 18F-FDG signals from the myocardium often preclude coronary artery imaging, despite attempts to suppress myocardial tracer uptake by dietary manipulation. These limitations of 18F-FDG for measuring changes in vascular inflammation arising from drug intervention highlight important unmet needs, which might be overcome by using a somatostatin receptor subtype-2 (SST2) PET tracer.

DETAILED DESCRIPTION:
Up-regulation of SST2 in activated macrophages represents a novel imaging target for measuring vascular inflammation, which has been previously examined in atherosclerosis using 68Ga-DOTATATE. To test the hypothesis that 68Ga-DOTATATE can quantify drug-induced changes in arterial inflammation, patients with primary hypercholesterolaemia (non-familial or familial) or mixed dyslipidaemia with stable cardiovascular Disease (CVD) and elevated LDL cholesterol ≥2.6 despite maximum tolerated statins with or without other lipid lowering therapies will undergo carotid artery 68Ga-DOTATATE PET-magnetic resonance imaging (MRI) in a randomised, double-blind, placebo-controlled study of inclisiran or colchicine.

In parallel, we will examine a novel method for detecting plaque composition based on analysis of ultrasound centre frequency shifts, which was developed by collaborators in Lund University, Sweden. The Ultrasound Plaque Structure Analysis (UPSA) method uses radiofrequency algorithms to create real-time tissue-like maps of carotid plaques. Participants in the study will undergo carotid ultrasound imaging using the UPSA method in addition to PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants >18 years old
* Able to give written, informed consent and to lie flat
* Have primary hypercholesterolaemia (non-familial or definite or possible heterozygous familial hypercholesterolaemia (HeFH) based on clinical criteria) or mixed dyslipidaemia, and
* History of CVD (acute coronary syndrome, coronary or other revascularisation procedures, coronary heart disease, ischaemic stroke, or peripheral arterial disease) and elevated LDL cholesterol ≥2.6 despite maximum tolerated statins with or without other lipid lowering therapies (see NICE TA 733), and
* Lipid lowering therapy unchanged for at least 6 weeks prior to screening, and
* Pre-existing carotid atherosclerotic plaque ≥15mm by B-mode ultrasound

Exclusion Criteria:

* Women of childbearing potential not using adequate contraception
* Contra-indication to MRI scanning
* Statin-associated myositis or liver function abnormality
* Already taking inclisiran or colchicine
* Sensitivity and/or contraindication to inclisiran or colchicine. Contraindications to colchicine include severe hepatic or renal impairment, blood disorders, and patients with renal or hepatic impairment who are taking a P-gp inhibitor or a strong CYP3A4 inhibitor
* Contrast allergy or contrast-nephropathy
* Chronic kidney disease (eGFR <30 mL/min/1.73 m2)
* Cardiovascular event within 6 months
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study
* Uncontrolled chronic inflammatory disorder
* History of recent malignancy deemed relevant to the study by the investigator
* Treatment with medications that result in significant drug to drug interactions with the study medications
* Current use of systemic corticosteroids or other immunosuppressive drugs
* Previous or planned carotid endarterectomy surgery or stenting on the index side

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Carotid 68Ga-DOTATATE PET | 12 weeks
  Relative change from baseline in carotid artery 68Ga-DOTATATE tissue-to-blood ratio in the index vessel
Carotid UPSA imaging | 12 weeks
  Relative change from baseline in carotid artery UPSA signal in the index vessel

SECONDARY OUTCOMES:
MRI plaque burden | 12 weeks
  Relative change from baseline in carotid artery total plaque burden and lipid-rich necrotic core measured by MRI
Carotid 68Ga-DOTATATE vs. serum lipids | 12 weeks
  Comparison of carotid 68Ga-DOTATATE imaging to serum lipids
Carotid 68Ga-DOTATATE vs. hsCRP | 12 weeks
  Comparison of carotid 68Ga-DOTATATE imaging to high-sensitivity C-reactive protein (hsCRP)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Tarkin, MBBS PhD, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306
- [Background] Pedersen SF, Sandholt BV, Keller SH, Hansen AE, Clemmensen AE, Sillesen H, Hojgaard L, Ripa RS, Kjaer A. 64Cu-DOTATATE PET/MRI for Detection of Activated Macrophages in Carotid Atherosclerotic Plaques: Studies in Patients Undergoing Endarterectomy. Arterioscler Thromb Vasc Biol. 2015 Jul;35(7):1696-703. doi: 10.1161/ATVBAHA.114.305067. Epub 2015 May 14. PMID 25977567